CLINICAL TRIAL: NCT03906682
Title: RAP Club: Improving Mental Health and School Performance in Urban Eighth Graders
Brief Title: Improving Mental Health and School Performance in Urban Eighth Graders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Institute of Education Sciences (U.S. Federal Agency); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: R305A160082-17; R01HD090022 (NIH)
Record Dates: First submitted 2018-11-14; First posted 2019-04-08 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Depressive Symptoms; Trauma, Psychological; Disruptive Behavior
Keywords: prevention; urban youth; mindfulness
MeSH Terms: conditions — Depression; Psychological Trauma; Problem Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAP Club program (Experimental): RAP Club is a 12-session universal prevention program delivered twice per week over six weeks during the school day. The program is delivered by a trained facilitator and young adult community member.
  Interventions: Behavioral: RAP Club
- Healthy Topics program (Active Comparator): Like RAP Club, Healthy Topics is a 12-session program delivered twice per week over six weeks during the school day. The program is delivered by a trained facilitator and young adult community member.
  Interventions: Behavioral: Healthy Topics

INTERVENTIONS:
Behavioral: RAP Club — RAP Club was adapted from a trauma treatment program called Structured Psychotherapy for Adolescents Responding to Chronic Stress (SPARCS). Core program components include psychoeducation, mindfulness, and cognitive-behavioral strategies.
  Arms: RAP Club program
Behavioral: Healthy Topics — Co-investigator Dr. Sibinga developed the Healthy Topics curriculum to function as an active control condition for randomized controlled trials in both clinic-based and school-based studies of mindfulness instruction for urban youth. Adapted from the Glencoe Health Curriculum (McGraw Hill), it was designed to control for the effects of a positive adult, time and attention, a small group learning environment, engaged instruction, and interesting material. The Healthy Topics curriculum has been successfully implemented as an effective active control condition, with student engagement and participation comparable to the intervention arm. The curriculum includes information about nutrition, exercise, sleep, drug use, and other topics related to physical health.
  Arms: Healthy Topics program

SUMMARY:
This study assesses: (1) the impact of the Relax, Be Aware, Do a Personal Rating (RAP) Club, a school-based prevention program for urban eighth graders, on students' emotional functioning and education outcomes; (2) potential moderators and mediators of RAP Club's effects; and (3) factors related to the implementation of RAP Club, including cost of delivery and perceptions of key stakeholders.

DETAILED DESCRIPTION:
Youth in low-income urban communities are often exposed to chronic stress and trauma, which poses risk for emotional, behavioral, and academic problems. This study will evaluate the impact of RAP Club, a trauma-informed school-based prevention program intended to promote positive emotional and academic development for eighth graders. Participants will be randomly assigned within schools to receive RAP Club or Healthy Topics, a health education active control condition.

The study will achieve the following specific aims:

1. Test whether students randomized to RAP Club have improved academic, social-emotional, and behavioral outcomes as compared to those randomized to Healthy Topics (e.g., student-reported mood and stress; teacher-rated academic performance; academic record data).
2. Explore potential moderators (e.g., baseline trauma exposure, emotional regulation) and mediators (e.g., changes in self-regulation and emotional symptoms) of RAP Club's effects.
3. Evaluate factors related to program implementation, including cost of delivering RAP Club versus Healthy Topics and perceptions of key stakeholders (teachers, group facilitators, students) regarding intervention acceptability and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Subject is attending eighth grade at a participating Baltimore City Public School
* Subject is not in a self-contained special education classroom
* Subject provides written parent permission and written assent

Exclusion Criteria:

* Non English-speaking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 615 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Teacher Rating of Social Competence Scale (TRSCS) | Past three weeks
  31-item teacher-rated scale of student classroom behavior using a 6-point Likert scale. Means are calculated for each subscale (Aggressive Behaviors, Oppositional Behavior, Attention and Concentration, Social and Emotional Competence). Higher scores reflect a higher level of that particular construct.
Strengths and Difficulties Questionnaire (SDQ) | Past 6 weeks
  Made up of 5 scales (Emotional Symptoms, Conduct Problems, Hyperactivity, Peer Problems, Prosocial Behavior). Several items (7, 21, 25, 11, and 14) are reverse coded. Total difficulties score is created by summing scores from all scales except the prosocial scale. The score ranges from 0-40 and is counted as missing if one of the 4 component scores is missing.
Academic Competence Evaluation Scale (ACES) | Past 6 weeks
  10-item teacher report of student academic functioning with 3 subscales (Engagement, Motivation, Academic Performance) that is rated on a 5-point Likert scale. Mean of items 1-9 provides the total score; subscales are calculated by taking the mean of relevant items. Higher scores indicate more academic competence.
Academic records | Past year
  Data on school performance collected by the 8th grade teacher as part of routine school practice.

SECONDARY OUTCOMES:
Child PTSD Symptom Scale Revised (CPSSR) | Past 2 weeks
  17-item self-report measure of trauma symptoms using a 4-point Likert scale. Items are summed to produce a total score. Higher scores indicate more trauma symptoms.
Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Symptoms | Past 7 days
  4-item self-report measure of anxiety symptoms using a 5-point Likert scale. Items are summed and then converted to standardized t score. Higher scores reflect higher frequency of anxiety symptoms.
Children's Depression Inventory - Short Form (CDI-S) | Past 2 weeks
  10-item self-report measure of depressive symptoms using a 5-point Likert scale. Items are summed to create a score ranging from 0-20; cutoffs can be used to determine depression severity. Higher scores reflect greater frequency of depression symptoms.
Youth Outcome Questionnaire Self-Report (YOQSR) | Past week
  64-item measure of youth psychological symptoms using a 5-point Likert scale. Items are summed to produce a total score, with higher scores indicating more psychological symptoms.
Brief Cope | Past 6 weeks
  28-item self-report measure of coping using a 4-point Likert scale. We intend to score this measure by using factor analysis to identify sub scales. In previous research, we have identified an adaptive subscale and maladaptive sub scale using this method. Higher scores indicate greater frequency of using a particular coping method.
Children's Response Style Questionnaire (CRSQ) | Past 6 weeks
  14-item self-report measure of rumination using a 4-point Likert scale. Mean score is calculated excluding item 14. Higher scores reflect greater tendency to engage in a ruminative response style.

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Mendelson, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The final study data will be computerized datasets that include demographic, behavioral, and emotional information. Data will be redacted to strip all subject identifiers. Datasets will be archived with The Inter-University Consortium for Political and Social Research (ICPSR) at the Institute for Social Research.
  ICPSR will provide: (1) data preparation tasks, which include reviewing data for confidentiality and usability, creation of a metadata record, generation of multiple data formats for dissemination and preservation, as well as assignment of a Digital Object Identifier (DOI); and (2) documentation to accompany the quantitative data including codebooks, variable and value labels for two quantitative data files containing up to 200 variables.
  A copy of the qualitative data with all identifying information redacted will be placed in ICPSR's data hosting service (openICPSR.org). A digital object identifier (DOI) will be issued for the files from this project.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After initial data analysis and preparation of major publications have been completed.
Access Criteria: Data files placed in the data hosting service are open access and freely available to the research community.
URL: https://www.icpsr.umich.edu/web/pages/